CLINICAL TRIAL: NCT04655846
Title: Efficacy of an Educational Intervention in Pregnant Adolescents for the Maintenance of Exclusive Breastfeeding
Brief Title: Efficacy of an Educational Intervention in Exclusive Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: lliana Ulloa Sabogal (Other)
Responsible Party: Sponsor-Investigator, lliana Ulloa Sabogal, Profesor, Universidad Industrial de Santander
Organization: Universidad Industrial de Santander (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2453
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Breastfeeding, Exclusive
Keywords: Breast Feeding; Education, Nursing; Pregnant Women; Adolescent
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Usual manage during prenatal control program
  Interventions: Behavioral: Nursing education about maternal care and usual education in maternity preparation course
- Intervention group (Experimental): Educational intervention towards the maintenance of exclusive breastfeeding in the first six months in first pregnant adolescents enrolled in the prenatal control program
  Interventions: Behavioral: Nursing intervention outcome: Breastfeeding Counseling (5244)

INTERVENTIONS:
Behavioral: Nursing intervention outcome: Breastfeeding Counseling (5244) — Educational sessions: The nursing professional will carry out 1 educational session per week, for 4 weeks; each lasting between 45 and 60 minutes. The topics that make up each of the activities are:
  1. Educational Session: Awareness towards the process of breastfeeding. Inform about the psychological and physiological benefits of breastfeeding.
  2. Educational session: Teach the composition of breast milk. Teach the baby's correct alignment, latch, and areolar understanding of the breast. Instruct on breastfeeding positions.
  3. Educational Session: Explain the extraction and conservation of breast milk.
  4. Educational session: Explain the signs, symptoms, and management strategies for duct obstruction, mastitis, and nipple trauma. Talk about your needs for rest, hydration, and diet during breastfeeding.
  Arms: Intervention group
Behavioral: Nursing education about maternal care and usual education in maternity preparation course — Educational intervention by a nursing professional on the provision of adequate care at the level of growth and development in infants under one year of age, activities not related to the breastfeeding process
  Arms: Control group

SUMMARY:
About 40% of children under six months are breastfed. However, in adolescent mothers there are greater barriers to making the decision to breastfeed. Counseling on breastfeeding could be a helpful intervention in sustaining this practice. This is a single-blind randomized controlled trial type study, with a control group that will receive routine care, and an intervention group that will additionally receive "Counseling: breastfeeding" through a maternity preparation course, both conducted by trained nurses. 59 pregnant women will be included in each group that attend the prenatal control program, for a total of 118 users. The level of knowledge about breastfeeding, the rate of cessation of breastfeeding and the rate of cessation will be evaluated in three measurements during follow-up.

DETAILED DESCRIPTION:
Introduction: The World Health Organization establishes that only 38% of children under six months of age in the developing world are exclusively breastfed and only 39% of children between 20 and 23 months they benefit from this practice. This problem is more evident in adolescent mothers, in whom the social, family and cultural influence, their level of knowledge, and the quality of health care services are decisive in the decision to give breast milk to their babies or not. sons. In this sense, nursing must design and implement educational intervention strategies for the promotion, protection and support of exclusive breastfeeding in the first six months of life.

Objective: To determine the efficacy of an educational intervention in first pregnant adolescents for the maintenance of exclusive breastfeeding in the first six months of life.

Methods: experimental study type randomized controlled clinical trial with first-pregnant adolescents assigned to an intervention group and a control group. The sample will be made up of a total of 118 first-pregnant women, 59 first-pregnant women in each study group.

The intervened group, in addition to receiving the usual prenatal care education, will receive an educational intervention of counseling on breastfeeding. The control group, in addition to the usual information on prenatal care, will receive an educational intervention related to infant care activities. The educational intervention will take place in 4 weekly sessions. Likewise, the intervention and control group will be given the final assessment of knowledge once the fourth educational intervention is finished and at 6 months postpartum. In addition, the maintenance of exclusive breastfeeding will be verified in the intervention and control group through home visits at two, four and six months postpartum.

Randomization: It will be carried out by blocks in groups of equal size, randomized 1: 1. The generation will be given by one of the researchers who will not perform the intervention, nor the initial or final evaluations.

Expected results: it is expected to increase the level of knowledge and a lower rate of abandonment of breastfeeding in the group of first pregnant adolescents operated on.

ELIGIBILITY:
Inclusion Criteria:

* First pregnant adolescents of Colombian nationality enrolled in the prenatal control program in three institutions of health
* First pregnant adolescents aged 14 years or older
* First pregnant adolescents with gestational age between 20 and 30 weeks
* Initial score less than or equal to 3.8 on the knowledge scale: Breastfeeding , described in the Nursing Results Classification

Exclusion Criteria:

* Pregnancy teenagers with psychiatric disorders and / or communication.
* Pregnant teenagers of Venezuelan nationality

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-12-18 (Estimated); Study Completion 2021-06-18 (Estimated)

PRIMARY OUTCOMES:
cessation rate of breastfeeding | 6 months
  The exclusive breastfeeding cessation rate during the first 6 months.

SECONDARY OUTCOMES:
Level of knowledge of breastfeeding process | 6 month
  The level of knowledge of the first pregnant adolescents about the breastfeeding process is evaluated through a questionnaire derived from the standardized outcome Knowledge: Breastfeeding (1800) of The Nursing Outcomes Classification (NOC) by Iowa University.
  This questionnaire consists of 7 indicators, with a Likert-type scale with a score from 1 to 5 (1: no knowledge, 2: little knowledge, 3: moderate knowledge, 4: substantial knowledge and 5: extensive knowledge) and the total score obtained goes from 7 to 35 points

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Industrial de Santander, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabogal IMU, Narino CCD, Monsalve MAM. Lactation counseling for maintaining exclusive breastfeeding in adolescent mothers: a trial protocol. Pilot Feasibility Stud. 2021 Dec 16;7(1):219. doi: 10.1186/s40814-021-00950-9. PMID 34915924